CLINICAL TRIAL: NCT03387917
Title: TLD-1, a Novel Liposomal Doxorubicin, in Patients With Advanced Solid Tumors: A Multicenter Open-label Single-arm Phase I Trial
Brief Title: TLD-1, a Novel Liposomal Doxorubicin, in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The premature termination is based on the unexpectedly low patient accrual to the clinical trial and the strategic considerations in the development of the TLD-1 after having included 13 out of 14 patients in the comparative PK part.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 65/16
Record Dates: First submitted 2017-11-21; First posted 2018-01-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; doxorubicin; TLD-1; phase I; Talidox; Liposomal
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: The trial uses an accelerated titration design (ATD) up to the occurrence of the first DLT, followed by a modified continual reassessment method (mCRM) for dose escalation part and randomized cross-over design for the comparative PK part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLD-1 (Experimental): Duration of treatment
  * 1 cycle: 21 days
  * 1 cycle: 28 days (only comparative PK part, in cycle 1 or 2)
  * until progression or occurrence of unacceptable toxicity or withdrawal, but
    * maximum 9 cycles for patients previously not treated with anthracyclines
    * maximum 6 cycles for patients previously treated with anthracyclines.
  * Dose: i.v., according to DL on day 1 of each cycle or tentative MTD
  Interventions: Drug: TLD-1
- Caelyx (only for comparative PK part) (Experimental): Duration of treatment
  * 1 cycle: 28 days
  * Caelyx is given only in one cycle (cycle 1 or 2)
  * Dose: i.v., 40mg/m2
  Interventions: Drug: Caelyx

INTERVENTIONS:
Drug: TLD-1 — TLD-1 is a new liposomal formulation of the anthracycline doxorubicin.
  Other Names: Talidox
  Arms: TLD-1
Drug: Caelyx — Caelyx is a liposomal formulation of the anthracycline doxorubicin
  Arms: Caelyx (only for comparative PK part)

SUMMARY:
TLD-1 is a novel liposomal formulation of doxorubicin (PEG surface) that compared favorably to conventional liposomal formulations of doxorubicin including Caelyx® in preclinical in vivo models. Particle features including size, charge distribution, lipid composition and drug release add up to a considerably altered particle behavior compared to Caelyx®, potentially explaining the lack of hand-foot-syndrome in respective animal models. Preclinical evaluation confirmed TLD-1 to be a promising new and innovative formulation of doxorubicin with promising activity and good tolerability.

DETAILED DESCRIPTION:
Despite impressive progress in the fields of surgical and immunological cancer therapies, most late-stage cancer treatments still heavily depend on conventional chemotherapeutics, which are often effective but also toxic, resulting in severe adverse effects limiting the dose and duration of therapy. Consequently, there remains a high unmet medical need for new innovative systemic treatments with an improved risk-benefit-profile.

Doxorubicin is a potent anthracycline used as a systemic treatment against several solid tumor including breast, ovarian and bladder cancer, small cell lung cancer and various types of sarcoma. However, Doxorubicin use is often limited due to hematological and non-hematological toxicity including cumulative cardiotoxicity with myocardial damage.

Cardiotoxicity has been substantially mitigated through the introduction of liposomal formulations such as Myocet and Caelyx/Doxil. Both products are associated with substantially lower rates of cardiac dysfunction during or post-treatment. Whereas Myocet's clinical use remains limited due to the intricate "bedside" reconstitution process, Caelyx has been associated with a high incidence of Palmar-Plantar Erythrodysesthesia (PPE) (also called hand-foot-syndrome), likely due to its long plasma half-life.

The development of TLD-1 (Talidox) aimed at combining the cardio-preserving properties of the liposomal delivery system with shorter blood circulation time in order to reduce the risk of PPE. Even though the pathophysiology of PPE is not yet fully understood, studies analyzing the correlation of dose and pharmacokinetic parameters with PLD toxic effects revealed that the severity of PPE correlated significantly with plasma half-life (t1/2).

Given its performance in preclinical trials, TLD-1 bears the potential for an improved benefit/risk profile compared to established liposomal doxorubicin formulations including Caelyx.

This first-in-human phase-I trial will evaluate the safety and will establish the maximal tolerated dose (MTD) and recommended phase II dose of TLD-1, and characterize specific dose limiting toxicities (DLT) of TLD-1. Moreover, the trial shall yield information on adverse events profile, pharmacokinetics and preliminary efficacy.

ELIGIBILITY:
Key inclusion criteria for dose escalation part:

* Final protocol until amendment 2: Patients with either histologically or cytologically confirmed advanced or recurrent solid tumor who failed standard therapy or for whom no effective standard therapy is available
* From Amendment 3 on: Patients with histologically or cytologically confirmed advanced malignant tumors of the breast, ovary, uterine or sarcoma who failed standard therapy or for whom no effective standard therapy is available.
* Patients may have received up to 3 prior lines of palliative systemic chemotherapy
* Patients with brain metastases must have undergone definitive treatment (surgery and/or radiation) at least 1 month prior to starting study drug and be documented as having stable disease by imaging and are on stable doses of steroids for at least 2 weeks.
* Adequate bone marrow, renal and hepatic function

Key inclusion criteria for comparative PK part:

* Patients with either histologically or cytologically confirmed advanced or recurrent breast or ovarian cancer of all histologies

  * Histologically-confirmed ovarian, fallopian tube or primary peritoneal cancer (collectively referred to herein as 'ovarian cancer') that is either platinum-resistant (disease progression within 6 months of the last receipt of platinum-based chemotherapy) or refractory (lack of response or disease progression while receiving the most recent platinum-based therapy).
  * Patients with ovarian cancer may have received up to 3 lines of prior cytotoxic chemotherapy, but maximum 1 of them in the platinumresistant/ refractory setting. Confirmed high-grade serous, endometrioid, or carcinosarcoma histotypes are permitted.
  * Patients with advanced or recurrent breast cancer may have received up to 2 prior lines of palliative cytotoxic chemotherapy.
* Patients with brain metastases must have undergone definitive treatment (surgery and/or radiation) at least 1 month prior to starting study drug and be documented as having stable disease by imaging and be on stable doses of steroids for at least 2 weeks.
* Adequate bone marrow, renal and hepatic function

Key exclusion criteria for dose escalation and comparative PK part:

* Significant cardiac disease or abnormality
* Patients who have received prior anthracyclines at a cumulative dose that exceeds 250mg/m2 for non-liposomal doxorubicin, 300mg/m2 for liposomal doxorubicin or 400mg/m2 for epirubicin and/or are refractory (during 3 months) to anthracyclines or have experienced allergic reactions or severe toxicity (grade 3 or 4) under anthracyclines
* Prior systemic chemotherapy/treatment for adjuvant/metastatic disease, radiotherapy, immunotherapy, or investigational agents within 28 days 5 half- life periods of previous therapy before registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | at 3 weeks
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: volume of distribution [Vd] | 2 months
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: Area under curve [AUC] | 2 months
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: Area under curve [Cmax] | 2 months
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: Terminal half life [t½] | 2 months
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: Clearance (CL) | 2 months
Descriptive pharmacokinetics (PK) of TLD-1 vs Caelyx: Ratio of unencapsulated to encapsulated drug over time for Caelyx and TLD-1 | 2 months

SECONDARY OUTCOMES:
Adverse Events (AEs) | at 7 months
Objective tumor response (OR) | at 7 months
Time to treatment failure (TTF) | at 7 months
Population pharmacokinetics (PK) of TLD-1: clearance (CL) | at 2 months
Population pharmacokinetics (PK) of TLD-1: volume of distribution (Vd) | at 2 months
Population pharmacokinetics: Area Under the Curve [AUC] | at 2 months
Population pharmacokinetics: Maximum Plasma Concentration [Cmax] | at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Hess, MD, Study Chair — Cantonal Hospital of St. Gallen; Anastasios Stathis, MD, Study Director — IOSI, Ospedale San Giovanni; Markus Jörger, Prof, Study Director — Cantonal Hospital of St. Gallen
Locations (5):
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur

REFERENCES:
- [Derived] Klose M, Colombo I, Gobat K, Koster KL, Haefliger S, Rabaglio M, Bastian S, Schwitter M, Zurrer-Hardi U, Eckhardt K, Hayoz S, Halbherr S, Sessa C, Michelet R, Mc Laughlin AM, Hess D, Stathis A, Kloft C, Joerger M. TLD-1, a Novel Liposomal Doxorubicin, in Patients with Solid Tumors: Comparative Pharmacokinetics and Final Results of a Multicenter Phase 1 Study (SAKK 65/16). Clin Pharmacokinet. 2025 Nov 18. doi: 10.1007/s40262-025-01588-z. Online ahead of print. PMID 41252081
- [Derived] Mc Laughlin AM, Hess D, Michelet R, Colombo I, Haefliger S, Bastian S, Rabaglio M, Schwitter M, Fischer S, Eckhardt K, Hayoz S, Kopp C, Klose M, Sessa C, Stathis A, Halbherr S, Huisinga W, Joerger M, Kloft C. Population pharmacokinetics of TLD-1, a novel liposomal doxorubicin, in a phase I trial. Cancer Chemother Pharmacol. 2024 Sep;94(3):349-360. doi: 10.1007/s00280-024-04679-z. Epub 2024 Jun 15. PMID 38878207
- [Derived] Colombo I, Koster KL, Holer L, Haefliger S, Rabaglio M, Bastian S, Schwitter M, Eckhardt K, Hayoz S, Mc Laughlin AM, Kloft C, Klose M, Halbherr S, Baumgartner C, Sessa C, Stathis A, Hess D, Joerger M. TLD-1, a novel liposomal doxorubicin, in patients with advanced solid tumors: Dose escalation and expansion part of a multicenter open-label phase I trial (SAKK 65/16). Eur J Cancer. 2024 Apr;201:113588. doi: 10.1016/j.ejca.2024.113588. Epub 2024 Feb 2. PMID 38377773